CLINICAL TRIAL: NCT00856947
Title: Vitamin D Supplementation During Pregnancy for Prevention of Asthma in Childhood: An Interventional Trial in the ABC (Asthma Begins in Childhood) Cohort
Brief Title: Vitamin D Supplementation During Pregnancy for Prevention of Asthma in Childhood
Acronym: ABCvitaminD
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Copenhagen Studies on Asthma in Childhood (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2008-007871-26
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Asthma
Keywords: wheeze; infections; allergy; eczema; vitamin D
MeSH Terms: conditions — Asthma; Respiratory Sounds; Infections; Hypersensitivity; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Active Comparator): Dietary supplement: 2400 IU Vitamin D3 (2 tablets of 1200 IU) from week 24 of gestation to 1 week after delivery
  Interventions: Dietary Supplement: Cholecalciferol D3
- Placebo (Placebo Comparator): Placebo: 2 placebo tablets with no active substance, identical to the active tablets, from week 24 of gestation to 1 week after delivery
  Interventions: Other: Placebo tablet

INTERVENTIONS:
Dietary Supplement: Cholecalciferol D3 — 2 tablets of 1200 IU daily from week 24 of gestation to 1 week after delivery
  Other Names: Vitamin D from Camette, Denmark
  Arms: Vitamin D
Other: Placebo tablet — 2 tablets containing no active substance
  Other Names: Placebo tablets from Camette, Denmark
  Arms: Placebo

SUMMARY:
The aim of this study is to prevent asthma symptoms (recurrent wheeze) in childhood by supplementation with high dose vitamin D to the mother during pregnancy. Participants are mothers and children of the ABC (Asthma Begins in Childhood) cohort. Mothers are recruited during pregnancy and receive daily supplement with 2400 IU of Vitamin D3 or placebo from week 24 og gestation to 1 week after delivery. In addition all mothers are advised to take the recommended dose of 400 IU vitamin D daily. The mothers in ABC also participate in an interventional trial with fish oil supplementation, and the vitamin D randomization is stratified by fish oil treatment group. The child is followed with acute and planned vits at the research unit, and wheeze is diagnosed according to predefined algorithms.

ELIGIBILITY:
Inclusion Criteria:

Mother:

* Pregnant in week 22-26 of gestation
* Participating in the ABC-cohort
* Living in Sealand, Denmark
* Fluent in Danish
* Willing to let the child participate in the study

Exclusion Criteria:

Mother:

* Intake of more than 400 IU of vitamin D during the last 6 months
* Endocrinological disease such as calcium metabolic disorder, parathyroid disorder, thyroid disorder or Diabetes type 1
* Tuberculosis
* Sarcoidosis
* In need of diuretics or heart medication including calcium channel blockers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2009-03; Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Persistent wheeze | 0 to 3 years of age
  Age at onset of persistent wheeze diagnosed according to predefined algorithm of recurrent troublesome lung symptoms, response to treatment and relapse after withdrawal of treatment

SECONDARY OUTCOMES:
Infections | 0 to 3 years of age
  Main analysis:
  • Number of lower respiratory tract infections registered in daily diaries
  Secondary analyses:
  * Acute otitis media
  * Number of upper respiratory tract infections
  * Number of other infections
  * Total number of infections
Allergic sensitization | 6 and 18 months of age
  Allergic sensitization at 6 and/or 18 months assessed by skin prick test and specific IgE in blood
Eczema | 0 to 3 years of age
  Age at onset of eczema diagnosed prospectively by research doctors according to predefined algorithm based upon Hanifin and Rajka criteria
Mothers levels of 25-OH-Vitamin D, PTH, Calcium, alkaline phosphatase | 1 week after delivery
Growth | 0 to 3 years of age
Asthma exacerbations | 0 to 3 years of age
  Age at onset of severe asthma exacerbation diagnosed by predefined criteria of acute severe asthma requiring oral/high dose inhaled steroids or acute hospital contact
Neurological development | 0-3 years
  Main analysis:
  • Cognitive development assessed at 2½ years using the cognitive part of Bayley Scales of Infant and Toddler Development, third edition
  Secondary analyses:
  * Milestone development monitored prospectively by the parents using a registration form based on The Denver Development Index and WHO milestones registration (combined assessment by principal component analysis)
  * Language development assessed at 1 and 2 years of age with the Danish version of The MacArthur Bates Communicative Developmental Inventory (CDI)
  * The child´s general development (language, fine and gross motor, social and problem solving) at 3 years of age assessed with Ages and stages Questioner, third edition (ASQ-3)
Growth | 0-3 years
  Main analysis:
  • Body composition (fat mass and bone mineral density) assessed by DEXA scan at 3 years of age
  Secondary analysis
  • Development of BMI from birth to 3 years assesses longitudinally in the research clinic
Systemic immune status | 18 months
  Main analysis Immune status at 18 months measured in stimulated whole blood as cytokine release (combined assessments by prinicipal component analyses)
  Secondary analyses Composition of immune cell subsets in whole blood at birth and at 18 months of age
Airway mucosal immune status | 4 weeks and 2 years
  Immune status measured in airway mucosal lining fluid at 4 weeks and 2 years of age (combined assessments by prinicipal component analyses for each age point)
17q21 genotype and sphingolipid metabolites | 6 months
  In a secondary analyses, we will determine the effect of 17q21 genotype on the efficacy of vitamin D supplementation in the prevention of asthma/wheeze. We will compute hazard ratios for the reduction in asthma/wheeze risk associated with prenatal supplementation, stratified by rs12936231. rs12936231 is a functional SNP influencing expression of ORMDL3, and given the role of ORMDL3 as a key sphingolipid biosynthesis regulator, we will subsequently investigate the relative abundance of sphingolipids between those in the vitamin D Intervention arm and those in the placebo group, stratified by 17q21 genotype. Finally we will identify interactions between prenatal vitamin D supplementation, rs12936231 genotype and sphingolipid metabolism in the risk of asthma/wheeze by age three.
Dental health | 6 year
  Caries and enamel defects (molar incisor hypomineralization, MIH) determined at a dental examination at age 6 years.

OTHER OUTCOMES:
Asthma | 3-10 years of age
  Asthma diagnosed from age 3 to 10 years based on the same predefined algorithm of recurrent troublesome lung symptoms, response to treatment after withdrawal of treatment, which was used for persistent wheeze at age 0-3 in phase 1 of the study. Primary outcome in phase 2 is current asthma at specific visits till age 10 years, which is diagnosed in children fulfilling the persistent wheeze algorithm at any point during the first 10 years of life and still needing inhaled corticosteroids at specific visits (3, 4, 5, 6, 8 and 10 years of age) to control the symptoms.
Lung function measurements | 5-10 years of age
  Spirometry measuring airflow assessed by FEV1, MMEF and FEV1/FVC ratio at age 5, 6, 8 and 10 years.
Infections | 3-10 years of age
  Prescribed medicine for infections. Types and length of infections
Growth | 3- 10 years of age
  Anthropometrics:
  Clinical follow up on the development of weight in kg (calibrated digital weight scales), height in cm (Harpenden stadiometer), waist-, thorax- and head circumference in cm (using tape; 3 times each) at every visit till age 10 years assessed longitudinally in the research clinic.
Eczema | 3-10 years of age
  Age at onset of eczema diagnosed prospectively by research doctors according to predefined algorithm based upon Hanifin and Rajka criteria
Allergic sensitization/atopy | 6-10 years of age
  Allergic sensitization at 6 and 10 years of age assessed by skin prick test (ALK-Abelló, Denmark) and specific IgE in blood (ImmunoCAP, PHarmacia Diagnostics AB, Sweden).
Airway mucosal immune status | 3-10 years of age
  Immune status measured in airway mucosal lining fluid at 3, 6 and 10 years of age (combined assessments by principal component analyses for each age point).
The diagnose allergic rhinitis | 3-10 years of age
  Allergic rhinitis will be diagnosed by combining allergic sensitization with symptom recording of troublesome congestion or sneezing or runny nose upon relevant exposure to allergens at age 3, 4, 5, 6, 8 and 10 years.
Asthma exacerbations: | 3-10 years of age
  Age at onset and number of severe asthma exacerbation diagnosed by predefined criteria of acute severe asthma requiring oral/ high dose inhaled steroids or acute hospital contact
Airway resistance | 3-10 years of age
  Measured by plethysmography (sRaw) at age 3, 4, 5, 6, 8 and 10 years.
Airway resistance | 3-5 years of age
  Multiple breath wash-out using SF6 and N2 as inert gasses to determined LCI, Scond and Sacin at ages 3, 4 and 5 years.
Bronchial reactivity: | at 6 years of age
  Provocative dose of methacholine leading to a 20% drop in FEV1 from baseline (PD20 value) at age 6 years.
Body composition | 3-13 years of age
  Body composition measured as fat mass, lean mass, bone mineral content (BMC) and bone mineral density assessed (BMD) through DXA scans at 3, 6 and years of age.
  Body impedance measurements at 10 years of age.
Airway inflammation: | 6-10 years of age
  Measurement of fractional exhaled nitric oxide (FeNO) at age 6, 8 and 10 years
Cognitive function | 10 years of age
  A 2,5 hours cognitive evaluation at 10 years of age. Cognitive functions from a broad spectrum of cognitive domains will be assessed with subtests both using paper pencil tests and Cambridge Neuropsychological Test Automated Battery .
MRI scanning of the Brain | 10 years of age
  MRI scanning of the Brain
Behavioral and psychopathological dimensions. | 6- 10 years of age
  Questionnaires will be administered to the parents.
Behavioral and psychopathological dimensions. | 10 years of age
  Behavioral and psychopathological dimensions will be assessed at 10 years of age.
  The childrens' potential psychiatric diagnoses will be ascertained through the semi-structured clinical interview Schedule for Affective Disorders and Schizophrenia for School-Age Children - Present and Lifetime Version (K-SADS-PL) first with a parent and next with the child.
Strength and Difficulties Questionnaire (SDQ)- Questionnaires | 6, 8 and 10 years of age
  The Strengths and Difficulties Questionnaire (SDQ) is a brief behavioural screening questionnaire about 3-16 year olds. Questionnaires will be administered to the parents to obtain their evaluation of their child's potential psychopathology and behavior problems. Scores will be calculated form the questionnaires in order validated methods
ADHD- RS- Questionnaires | 8 and 10 years of age
  The ADHD Rating Scale obtains parent ratings regarding the frequency of each ADHD symptom based on DSM criteria.
  Questionnaires will be administered to the parents to obtain their evaluation of their child's potential psychopathology and behavior problems. Scores will be calculated form the questionnaires. Scores will be calculated form the questionnaires in order validated methods.
Social Responsive Scale, Second version (SRS-2) | 10 years of age
  The SRS-2 identifies social impairment associated with autism spectrum disorders (ASDs) and quantifies its severity Questionnaires will be administered to the parents to obtain their evaluation of their child's potential psychopathology. Scores will be calculated form the questionnaires. Scores will be calculated form the questionnaires in order validated methods.
The Child Behavior Checklist school-age version (CBCL) | 10 years of age
  The Child Behavior Checklist (CBCL) is a widely used questionnaire to assess behavioral and emotional problems.
  Questionnaires will be administered to the parents to obtain their evaluation of their child's potential psychopathology and behavior problems. Scores will be calculated form the questionnaires. Scores will be calculated form the questionnaires in order validated methods.
The Behavior Rating Inventory of Executive Function 2nd edition (BRIEF-2) | 10 years of age
  The BRIEF-2 is a set of questionnaires for parents and teachers , designed to evaluate executive function from multiple perspectives.
  Questionnaires will be administered to the parents to obtain their evaluation of their child's potential psychopathology. Scores will be calculated form the questionnaires. Scores will be calculated form the questionnaires in order validated methods.
Bone fractures | 0-13 years of age
  Description: Assessed by medical record checks including all radiologically verified fractures of larger long bones (i.e. clavicle, radius, ulna, tibia, fibula, femur and humerus). Outcome analyses: total no. of fractures age 0-13 years.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Bønnelykke, MD, PhD, Principal Investigator — Copenhagen Studies on Asthma in Childhood
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital of Copenhagen, Gentofte Municipality, Gentofte
  - Næstved Hospital, Pediatric Department, Næstved, Næstved

REFERENCES:
- [Derived] Palacios C, Kostiuk LL, Cuthbert A, Weeks J. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2024 Jul 30;7(7):CD008873. doi: 10.1002/14651858.CD008873.pub5. PMID 39077939
- [Derived] Aagaard K, Mollegaard Jepsen JR, Sevelsted A, Horner D, Vinding R, Rosenberg JB, Brustad N, Eliasen A, Mohammadzadeh P, Folsgaard N, Hernandez-Lorca M, Fagerlund B, Glenthoj BY, Rasmussen MA, Bilenberg N, Stokholm J, Bonnelykke K, Ebdrup BH, Chawes B. High-dose vitamin D3 supplementation in pregnancy and risk of neurodevelopmental disorders in the children at age 10: A randomized clinical trial. Am J Clin Nutr. 2024 Feb;119(2):362-370. doi: 10.1016/j.ajcnut.2023.12.002. Epub 2023 Dec 9. PMID 38072183
- [Derived] Brustad N, Yang L, Chawes BL, Stokholm J, Gurdeniz G, Bonnelykke K, Bisgaard H. Fish Oil and Vitamin D Supplementations in Pregnancy Protect Against Childhood Croup. J Allergy Clin Immunol Pract. 2023 Jan;11(1):315-321. doi: 10.1016/j.jaip.2022.09.027. Epub 2022 Sep 30. PMID 36184023
- [Derived] Mohammadzadeh P, Rosenberg JB, Vinding R, Mollegaard Jepsen JR, Lindberg U, Folsgaard N, Erlang Sorensen M, Sulaiman D, Bilenberg N, Mitta Raghava J, Fagerlund B, Vestergaard M, Pantelis C, Stokholm J, Chawes B, Larsson H, Glenthoj BY, Bonnelykke K, Ebdrup BH, Bisgaard H. Effects of prenatal nutrient supplementation and early life exposures on neurodevelopment at age 10: a randomised controlled trial - the COPSYCH study protocol. BMJ Open. 2022 Feb 1;12(2):e047706. doi: 10.1136/bmjopen-2020-047706. PMID 35105560
- [Derived] Knihtila HM, Kelly RS, Brustad N, Huang M, Kachroo P, Chawes BL, Stokholm J, Bonnelykke K, Pedersen CT, Bisgaard H, Litonjua AA, Lasky-Su JA, Weiss ST. Maternal 17q21 genotype influences prenatal vitamin D effects on offspring asthma/recurrent wheeze. Eur Respir J. 2021 Sep 23;58(3):2002012. doi: 10.1183/13993003.02012-2020. Print 2021 Sep. PMID 33653805
- [Derived] Sass L, Vinding RK, Stokholm J, Bjarnadottir E, Noergaard S, Thorsen J, Sunde RB, McGrath J, Bonnelykke K, Chawes B, Bisgaard H. High-Dose Vitamin D Supplementation in Pregnancy and Neurodevelopment in Childhood: A Prespecified Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2020 Dec 1;3(12):e2026018. doi: 10.1001/jamanetworkopen.2020.26018. PMID 33289844
- [Derived] Brustad N, Garland J, Thorsen J, Sevelsted A, Krakauer M, Vinding RK, Stokholm J, Bonnelykke K, Bisgaard H, Chawes BL. Effect of High-Dose vs Standard-Dose Vitamin D Supplementation in Pregnancy on Bone Mineralization in Offspring Until Age 6 Years: A Prespecified Secondary Analysis of a Double-Blinded, Randomized Clinical Trial. JAMA Pediatr. 2020 May 1;174(5):419-427. doi: 10.1001/jamapediatrics.2019.6083. PMID 32091548
- [Derived] Norrisgaard PE, Haubek D, Kuhnisch J, Chawes BL, Stokholm J, Bonnelykke K, Bisgaard H. Association of High-Dose Vitamin D Supplementation During Pregnancy With the Risk of Enamel Defects in Offspring: A 6-Year Follow-up of a Randomized Clinical Trial. JAMA Pediatr. 2019 Oct 1;173(10):924-930. doi: 10.1001/jamapediatrics.2019.2545. PMID 31381020
- [Derived] Wolsk HM, Chawes BL, Litonjua AA, Hollis BW, Waage J, Stokholm J, Bonnelykke K, Bisgaard H, Weiss ST. Prenatal vitamin D supplementation reduces risk of asthma/recurrent wheeze in early childhood: A combined analysis of two randomized controlled trials. PLoS One. 2017 Oct 27;12(10):e0186657. doi: 10.1371/journal.pone.0186657. eCollection 2017. PMID 29077711
- [Derived] Chawes BL, Bonnelykke K, Stokholm J, Vissing NH, Bjarnadottir E, Schoos AM, Wolsk HM, Pedersen TM, Vinding RK, Thorsteinsdottir S, Arianto L, Hallas HW, Heickendorff L, Brix S, Rasmussen MA, Bisgaard H. Effect of Vitamin D3 Supplementation During Pregnancy on Risk of Persistent Wheeze in the Offspring: A Randomized Clinical Trial. JAMA. 2016 Jan 26;315(4):353-61. doi: 10.1001/jama.2015.18318. PMID 26813208